CLINICAL TRIAL: NCT05454397
Title: A Study on the Status of Nutritional Risk Screening and Nutritional Therapy in Neurology Hospitalized Stroke Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: First Affiliated Hospital of Fujian Medical University (Other); Yantai Yuhuangding Hospital (Other); The First Hospital of Jilin University (Other); Qilu Hospital of Shandong University (Other); ZHEJIANG PROVINCE XIAOSHAN HOSPITAL (Unknown); Affiliated Wenling Hospital of Wenzhou Medical University (Other); Ganzhou People's Hospital (Unknown); Affiliated Hospital of Jining Medical hospital (Unknown); Henan Provincial People's Hospital (Other); Zhongda Hospital (Other); The Second Affiliated Hospital of Harbin Medical University (Other); The First People's Hospital of Kunshan (Other); The 2nd Affiliated Hospital of Wenzhou Medical University (Unknown); THE FIRST PEOPLE'S HOSPITAL OF JIASHAN (Unknown); First Affiliated Hospital Xi'an Jiaotong University (Other); Fujian Province Zhangzhou Hospital (Unknown); People's Hospital of Chongqing (Other); Nanjing Zijin Hospital (Unknown); Red Cross Hospital, Hangzhou, China (Other); Wenzhou Hospital of Chinese Medicine (Unknown); Kaifeng Central Hospital (Other); First Affiliated Hospital of Guangxi Medical University (Other); Zhongshan Hospital of Xiamen University (Unknown); Xi'an Encephalopathy of Traditional Chinese Medicine Hospital (Unknown); 903 Hospital of Chinese People's Liberation Army (Other); Xiangya Hospital of Central South University (Other); Second Affiliated Hospital of Suzhou University (Other); Tongji Hospital (Other); The Affiliated Hospital o fQingdao University (Unknown); The First Affiliated Hospital of Anhui Medical University (Other); Yancheng Third People's Hospital (Unknown); Linyi People's Hospital (Other); Dongfang Hospital Beijing University of Chinese Medicine (Other); The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2020-234
Record Dates: First submitted 2022-07-01; First posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2021-10

CONDITIONS: Acute Stroke
Keywords: Stroke; Dysphagia;Nutrition management；
MeSH Terms: conditions — Stroke | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- case group: Patients with acute stroke with nutritional risk
  Interventions: Other: Observational study, no intervention

INTERVENTIONS:
Other: Observational study, no intervention — Observational study, no intervention

SUMMARY:
Stroke is the leading cause of premature death and disability, and early recognition and treatment of dysphagia is fundamental to stroke management. Early and full tube feeding in the acute phase of stroke helps to address nutritional problems resulting from dysphagia and impaired consciousness and helps to reduce morbidity and mortality and poor outcomes. Current guidelines for acute stroke management do not address the goal of tube feeding of enteral nutrition for energy and protein. In the treatment of acute stroke, there is a strong global focus on pharmacological thrombolysis or mechanical thrombolysis, with nutritional interventions being a less explored topic. Real-world evidence on large samples, feeding attainment and outcomes, and nutrition in the acute phase of stroke is lacking in China . The aim of this study was to understand the current status of nutritional therapy in stroke hospitalization in neurology and its impact on prognosis nationwide, and to improve the standardized management process of enteral nutrition therapy in the acute phase of stroke.

DETAILED DESCRIPTION:
Malnutrition is a common geriatric syndrome with a disproportionate incidence in geriatric and neurology inpatients. In recent years, national nutritional surveys of geriatric inpatients have shown that about 2/3 of geriatric inpatients have nutritional problems; only half of neurology inpatients at high risk receive nutritional support, and inadequate nutrition exacerbates primary disease, increases complications, makes hospital stays longer, and ultimately affects patient survival outcomes.

To increase comprehensive and up-to-date research on the current status of nutritional therapy in geriatric and neurology inpatients, and to lay the foundation for future standardized treatment and standardized management, we conducted a nationwide survey on the current status of nutritional risk screening and treatment in geriatric and neurology inpatients. The aim is to raise the level of clinicians' awareness of malnutrition and nutritional risk in hospitalized patients, standardize clinical practice, and properly implement nutritional support to improve patients' clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Newly admitted stroke patients admitted to neurology, age ≥18 years, within 7 days of onset, expected survival >3 months (i.e., not end-stage), expected neurology stay 7-10 days；
* At risk of malnutrition (MUST ≥ 2 points) or at nutritional risk (NRS2002 ≥ 3 points), sign an informed notice.

Exclusion Criteria:

* Transferred during treatment, contraindications to nutritional therapy (e.g., hemodynamic instability, gastrointestinal bleeding (bleeding >100 ml), other nutritional studies, pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly admitted stroke patients admitted to the neurology unit, ≥18 years of age, within 7 days of onset, expected survival >3 months, expected neurology stay 7-10 days, and at risk of malnutrition (MUST ≥2 points) or at nutritional risk (NRS2002 ≥3 points). Patients' age, sex, hospital, hospitalization number, height, primary diagnosis on admission, and previous underlying disease were collected.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2022-10-15 (Estimated); Study Completion 2023-10-15 (Estimated)

PRIMARY OUTCOMES:
Nutrition implementation rate | The first day of admission； the seventh day of admission； the day before discharge.
  Proportion of patients hospitalized for stroke who were given nutritional support
Nutrition compliance rate of stroke inpatients | The first day of admission； the seventh day of admission； the day before discharge.
  Percentage of patients hospitalized for stroke whose nutritional indicators and nutritional status met the guidelines after being given nutritional support

SECONDARY OUTCOMES:
30-day post-discharge mortality | 30-day post-discharge
  Proportion of enrolled patients who died 30 days after discharge from the hospital
Infection rate | 30-day post-discharge
  Proportion of enrolled patients with pulmonary infection 30 days after discharge from hospital.
Readmission rate | 30-day post-discharge
  Proportion of patients enrolled who were readmitted for various reasons 30 days after discharge.
Functional prognosis | 30-day post-discharge
  Functional prognosis of the enrolled patients, such as life skills, motor and sensory functions, cognitive functions and swallowing functions.

CONTACTS AND LOCATIONS:
Overall Officials: Suyue Pan, M.D., Ph.D., Principal Investigator — Department of Neurology, Nanfang Hospital, Southern Medical University
Locations (34):
- China (34):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Dongfang Hospital of Beijing University of Chinese Medicine, Beijing, Beijing Municipality
  - The First Afilliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - Fujian Province Zhangzhou Hospital, Zhengzhou, Fujian
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Kaifeng Central Hospital, Kaifeng, Henan
  - Henan Provincial People'S Hospital, Zhengzhou, Henan
  - Tongji Hospital of Tongji Medical College of HUST, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The First People'S Hospital of Kunshan, Kunshan, Jiangsu
  - Nanjing Zijin Hospital, Nanjing, Jiangsu
  - Zhongda Hospital Southeast Universtiy, Nanjing, Jiangsu
  - The second Affiliated Hospital of Suzhou University, Suzhou, Jiangsu
  - Yancheng Third People's Hospital, Yancheng, Jiangsu
  - Ganzhou People'S Hospital, Ganzhou, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Affiliated Hospital of Jining Medical Hospital, Jining, Shandong
  - Linyi People'S Hospital, Linyi, Shandong
  - Qilu Hospital of Shandong University(Qingdao), Qingdao, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Xi'an Encephalopathy of Traditional Chinese Medicine Hospital, Xi’an, Shanxi
  - Chongqing People's Hospital, Chongqing, Sichuang
  - Red Cross Hospital of Hangzhou, Hangzhou, Zhejiang
  - Zhejiang Province Xiaoshan Hospital, Hanzhou, Zhejiang
  - The First People'S Hospital of Jiashan, Jiaxing, Zhejiang
  - The First People'S Hospital of Wenling, Wenling, Zhejiang
  - The 2nd Affiliated Hospital and Yuying Children's Hospital of WMU, Wenzhou, Zhejiang
  - Wenzhou Hospital of Chinese Medicine, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No